CLINICAL TRIAL: NCT04351945
Title: A Study of Endocrine Changes and Their Correction in Heart and Lung Transplant Recipients and Donors
Brief Title: Endocrine Changes and Their Correction in Heart and Lung Transplant Recipients and Donors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Principal Investigator, Andrea Szekely, professor, Semmelweis University Heart and Vascular Center
Other Study IDs: VSZÉK TRANSPLANT
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Endocrine System Diseases; Thyroid Diseases; Cortisol Deficiency; Diabetes Insipidus; End-stage Heart Failure; End Stage Lung Disease
Keywords: transplantation; endocrine
MeSH Terms: conditions — Endocrine System Diseases; Thyroid Diseases; Diabetes Insipidus | interventions — Hematologic Tests; Transplantation; Device Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood test: Patients will have a blood test to define hormone levels.
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Hormone levels will be measured just before transplantation, and three day after the transplantation. In case of the donors hormone levels will be defined during the explantation.
  Other Names: transplantation; explantation

SUMMARY:
The aim of this study is to assess the impact of endocrine changes and their correction on survival and organ function in heart and lung transplant recipients. This study also features an investigation of the hormone levels and hormonal replacement therapy of the donors to study its role in the function of the transplanted hearts and lungs.

Thyroid hormones (TSH, thyroxine, tri-iodothyronine), cortisol and the antidiuretic hormone will be studied.

The former two hormone levels will be defined in the recipients just before transplantation and three days later. In the case of the donors all three hormones will be recorded at the time of the explantation. The investigators would like to record the hormonal replacement therapy in all our patients as well to see it's effect on survival and on the transplanted organ function.

After the transplantation during the hospital stays all the important hemodynamic parameters, laboratory parameters, the result of the medical imagings, the medication, the length of ICU and hospital stay and the complications were recorded.

Recipients will be followed for five years. Organ function will be assessed every three month for a year, after than every six month for further four years. Investigator would like to record the result of the cardiac echocardiography, spirometries, imaging, and complications. Our purpose is to compare these results against the endocrine disorders and the replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age admitted for heart or lung transplantation and their organ donors.
* written consent from the recipients

Exclusion Criteria:

* lack of consent
* non-evaluable patient due to insufficient clinical information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart or lung transplation and their organ donors.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The composite of in-hospital death of any cause | Patient will be followed during the hospital stay, an expected average of a month.
  In-hospital death of any cause
Endocrine changes and their correction in heart and lung tranplant recipients | 5 years
  Five year mortality rate
Endocrine changes and their correction in heart and lung tranplant donors | one month
  Number of successfully transplanted organs

SECONDARY OUTCOMES:
Endocrine changes and their correction in heart tranplant recipients | five years
  The function of the transplanted heart
Endocrine changes and their correction in lung tranplant recipients | five years
  The function of the transplanted lung
Evidence of clinically definite postoperative complications | five years
  Complications occuring during five year after the transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Andrea dr. Székely, MD PhD, Study Director — Semmelweis University; Ágnes dr. Sándor, MD, Principal Investigator — Semmeweis University; András dr. Szabó, MD, Principal Investigator — Semmelweis University
Locations (1):
- Heart and Vascular Center, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No